CLINICAL TRIAL: NCT04728035
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Irinotecan Liposome Injection in Patients With Advanced Breast Cancer
Brief Title: Study of Irinotecan Liposome Injection in Patients With Advanced Breast Cance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE072-CSP-002
Record Dates: First submitted 2021-01-18; First posted 2021-01-28 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2020-12

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation (part 1) (Experimental): Patients will receive irinotecan liposome injection (CSPC) at the initial starting dose until progression or unacceptable toxicity.
  Interventions: Drug: Irinotecan Liposome Injection
- Dose expansion (part 2) (Experimental): Once the appropriate dose has been established in Part 1, patients will be enrolled into two expansion cohorts according to the sub-type of breast cancer.
  Interventions: Drug: Irinotecan Liposome Injection

INTERVENTIONS:
Drug: Irinotecan Liposome Injection — Irinotecan Liposome Injection

SUMMARY:
This study is an open-label, single-arm, phase I study of irinotecan liposome injection in patients with advanced breast cancer. The purpose of this study is to evaluate the safety, efficacy and pharmacokinetics of irinotecan liposome injection in patients with advanced breast cancer.

DETAILED DESCRIPTION:
This is an open-label, single-arm, phase I study with a dose-escalation phase (part 1) and a dose-expansion phase (part 2). In part 1, patients will receive irinotecan liposome injection (CSPC) at the initial starting dose until progression or unacceptable toxicity. Dosages will be escalated by certain increments in subsequent cohorts. Once the appropriate dose has been established in part 1, patients will be enrolled into two expansion cohorts in part 2.

ELIGIBILITY:
Inclusion Criteria:

All patients 1.Female aged between 18 and 75 years.

2.Histologically or cytologically confirmed breast cancer.

3.At least one measurable lesion according to RECIST 1.1.

4.The time interval between the end of the last anti-tumor treatment and the first administration of irinotecan liposome injection is restricted as follows:

(1) More than 6 weeks for nitrosoureas (such as carmustine, lomustine, etc.) or mitomycin C.

(2) More than 3 weeks for cytotoxic chemotherapeutics, immunotherapy such as PD-1/PD-L1 and biotherapy.

(3) More than 2 weeks (five half-lives, whichever is longer) for oral fluorouracil, oral small molecule targeted drugs, and endocrine therapy.

(4) More than 2 weeks for Radiotherapy. (5) More than 2 Weeks for traditional Chinese medicine with anti-tumor indications.

5.Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.

6.Life expectancy >3 months.

7.Patient should not receive blood transfusion or supportive care (eg. EPO, G-CSF or others) within 14 days before the initiate dose, and laboratory test should meet the following criteria: neutrophile count ≥1.5×10^9/L platelet count ≥100×10^9/L hemoglobin ≥90 g/L or ≥5.6 mmol/L serum creatinine ≤1.5×ULN and creatinine clearance rate ≥50 mL/min total bilirubin ≤1×ULN AST and ALT ≤2.5×ULN

8.Patient with reproductive potential must agree to use adequate contraception from the signing of informed consent to at least 6 months after the trial completion and have a negative serum pregnancy test within 7 days before enrollment.

9.Ability to understand and the willingness to sign a written informed consent.

Additional criteria for dose escalation and cohort 1 in dose expansion

1.Meet the molecular classification criteria for triple-negative breast cancer.

2.Patients with locally recurrent or metastatic disease who have received at least two prior chemotherapeutic regimens for breast cancer and had failed to prior chemotherapy due to progression or intolerable toxicity:

(1)Early neoadjuvant or adjuvant chemotherapy for localized disease that progresses to unresectable locally advanced or metastatic disease within 12 months after completion is one of the permitted previous chemotherapy regimens.

(2)PARP inhibitor for patients with germline BRCA1/BRCA2 mutations who have been treated with approved PARP inhibitors, is one of the permitted prior chemotherapy regimens.

3.Previous treatment with taxanes and anthracyclines was required regardless of the stage of disease (neoadjuvant, adjuvant or palliative). Those who have contraindications or intolerance to a certain drug above should receive at least one cycle of treatment with this drug, and can be exempted from the requirements for the use of this drug.

Additional criteria for cohort 2 in dose expansion

1.HER2 negative breast cancer defined as 0 - 1+ by immunohistochemistry or FISH negative result.

2.Evidence of new and/or progressive brain metastases following previous radiotherapy (WBRT and/or SRS and/or gamma knife) and/or surgery.

3.At least one measurable brain lesion (≥10 mm on T1-weighted, gadolinium-enhanced magnetic resonance imaging).

Exclusion Criteria

1. Patients who have received any investigational drug within 4 weeks of the first dose of the study drug.
2. Patients who have undergone major organ surgery (excluding needle biopsy) or have significant trauma within 4 weeks prior to the first dose of the study drug, or have a schedule for major surgery during the trial.
3. Patients who have concomitant use of strong CYP3A4 inhibitors or inducers within 2 weeks prior to receiving the first dose of irinotecan liposome injection, or CYP3A4 inhibitors or UGT1A1 inhibitors within 1 week prior to receiving the first dose of irinotecan liposome injection, or those who could not suspend the above drugs during the study.
4. Patients who received systemic glucocorticoids (prednisone >10 mg/day or equivalent dose of the similar drugs) or other immunosuppressive agents within 14 days before the first dose of the study drug. Except for local, ocular, intra-articular, intranasal, and inhaled glucocorticoids, short term use of glucocorticoids for preventive treatment (e.g., prevention of contrast allergy). Cohort 2 in dose expansion is not limited.
5. Patients who have received prior topoisomerase I inhibitor treatment, including irinotecan or other investigational agents.
6. Known hypersensitivity (CTCAE 5.0≥3) to any of the components of irinotecan liposome injection, or other liposomal products.
7. Patients with central Nervous System (CNS) metastasis meet any of the following criteria: Cohort 2 in dose expansion is not limited.

(1)Patients who have developed new or progressive brain metastasis following cranial radiation or surgery.

(2)Patients with the symptomatic Central Nervous System (CNS) metastasis who have used cortisol, radiotherapy, dehydration drugs, etc. to control symptoms in the past two weeks.

(3)Patients with carcinomatous meningitis.

(4)Patients with brainstem (midbrain, pons, medulla oblongata) metastasis.

(5)Patients have other evidence indicates that the patient's central nervous system metastasis or meningeal metastasis has not been controlled and is judged unsuitable for enrollment by the investigator.

8.Patients who have pulmonary lymphatic dissemination and metastasis, leading to dyspnea at rest, may need to be combined with other treatments, such as oxygen inhalation, which is judged not suitable for enrollment by the investigator.

9.Prior radiation therapy encompassing more than 30% of bone marrow.

10.Patients have unresolved adverse reactions > grade 1 (CTCAE 5.0) from previous anti-tumor treatment (except for the peripheral neuropathy < grade 2, alopecia, and other toxicity judged no safety risk by investigators).

11.History of autoimmune disease, immunodeficiency (including HIV test positive), or other acquired or congenital immunodeficiency, or organ transplantation.

12.Patients with known Hepatitis B Virus (HBV DNA>2000 IU/ml), Hepatitis C Virus (anti-HCV positive), or other uncontrolled active infections.

13.Chronic gastrointestinal dysfunction with diarrhea as the main symptom, such as Crohn's disease, ulcerative colitis, malabsorption or Diarrhea ≥ grade 1, intestinal obstruction, or other gastrointestinal diseases of clinical significance as judged by the investigators.

14.Previous malignancies in the past five years (except basal cell carcinoma, squamous cell carcinoma, superficial bladder carcinoma, local prostate carcinoma, carcinoma in situ of cervical, or of others that have been radically resected and have not recurred).

15.History of serious cardiovascular disease, including but not limited to:

1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block, etc.
2. Patients with prolonged QT/QTc interval in baseline electrocardiogram (ECG) (QTcF > 480 ms, Fridericia formula: QTcF = QT/RR0.33, RR = 60/heart rate).
3. Patients with myocardial infarction, angina pectoris, coronary angioplasty or stent, deep vein thrombosis, stroke within 6 months before enrollment.
4. Baseline echocardiography (ECHO) or cardiac radionuclide scanning (MUGA) techniques showed left ventricular ejection fraction (LVEF) ≤ 50%, or NYHA grade Ⅲ and above.
5. Poorly controlled hypertension (systolic blood pressure≥150 mmHg and/or diastolic blood pressure≥ 95 mmHg with optimal treatment.
6. Previous or current cardiomyopathy.
7. Patients with clinically significant abnormal electrocardiogram (ECG)according to the investigator's assessment.

16. Uncontrolled third lacunar effusion, improper for enrollment by investigator's assessment.

17. Patients with alcohol or drug dependence.

18. Pregnant or lactating women.

19.History of explicit neurological or psychiatric disorders, including epilepsy or dementia.

20. Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration, or interfere with the interpretation of safety results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (AEs) and serious adverse events (SAEs) | Up to six months after the last patient's first administration
  The AEs and SAEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0.
Dose limiting toxicity (DLT) | Up to 28 days post-product injection
  DLT will be assessed according to NCICTCAE v5.0.
Maximum Tolerated Dose (MTD, if available) | Up to 28 days post-product injection
  MTD was defined as the previous dose level at which 2 out of 6 patients experienced a DLT.
Recommended Phase 2 Dose (RP2D) | Up to the end of the part 1
  RP2D was defined as the dose level chosen by the sponsor (in consultation with the investigators) for the dose expansion arms, based on safety, tolerability data collected during the dose escalation portion of the study.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to six months after the last patient's first administration
  The percentage of patients who achieve a complete response (CR) or partial response (PR) based on the modified Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
Progression-Free Survival (PFS) | Up to six months after the last patient's first administration
  Time from date of the first dose to date of recorded disease progression or death, whichever occurs first.
Disease Control Rate (DCR) | Up to six months after the last patient's first administration
  The percentage of patients who achieve a CR, PR or stable disease (SD) based on the modified RECIST 1.1.
Duration of Response (DOR) | Up to six months after the last patient's first administration
  Time from first documented response (CR or PR whichever occurs first, based on investigator's assessment using RECIST 1.1) to date of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to six months after the last patient's first administration
  Time from date of the first dose to date of death from any cause.
CNS objective response rate (CNS ORR) | Up to six months after the last patient's first administration
  The percentage of patients who achieve a CR or PR based on Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) in Cohort 2 of dose expansion.
CNS clinical benefit rate (CNS CBR) | Up to six months after the last patient's first administration
  The percentage of patients who achieve a CR, PR or SD based on RANO-BM in Cohort 2 of dose expansion.
The Area under the concentration-time curve from time zero to infinity (AUCinf) | -30minutes~168hours
  AUCinf of total irinotecan,wrapped irinotecan, free irinotecan and SN-38 will be measured for the test product .
The Maximum observed plasma concentration (Cmax) | -30 minutes~168 hours
  Cmax of total irinotecan，wrapped irinotecan, free irinotecan and SN-38 will be measured for the test product .
The terminal elimination half-life (T1/2) | -30 minutes~168 hours
  T1/2 of total irinotecan,wrapped irinotecan, free irinotecan and SN-38 will be measured for the test product.
The time to maximum concentration (Tmax) | -30minutes~168 hours
  Tmax of total irinotecan,wrapped irinotecan, free irinotecan and SN-38 will be measured for the test product .
The Apparent volume of distribution (Vd) | -30 minutes~168 hours
  Vd of total irinotecan will be measured for the test product.

OTHER OUTCOMES:
UGT1A1 gene polymorphism and Topoisomerase I (Topo I) expression | Up to six months after the last patient's first administration
  UGT1A1 gene polymorphism and Topoisomerase I (Topo I) expression

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hosptial of CAMS, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Fan Y, Zhang Q, Yan M, Qu X, Yin Y, Sun T, Yang J, Wang Y, Wang X, Niu Z, Wang X, Sun S, Zhao W, Liu Y, Niu M, Zhao X, Xu B. Intravenous liposomal irinotecan in metastatic triple-negative breast cancer after >/= 2 prior lines of chemotherapy: a phase Ib study. Nat Commun. 2025 Jan 2;16(1):3. doi: 10.1038/s41467-024-55090-4. PMID 39746964